CLINICAL TRIAL: NCT02005432
Title: Three Arm, Prospective, Single-blind, Randomized Study Comparing Ranibizumab Plus Green Diode Laser Versus Ranibizumab Plus Pattern Scan Laser (Pascal) Versus Ranibizumab (Monotherapy) for Proliferative Diabetic Retinopathy.
Brief Title: PASCAL Laser Versus ETDRS Laser Associated With Intravitreal Ranibizumab (IVR) Versus Only IVR for Proliferative Diabetic Retinopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rafael de Montier P. Barroso, MD, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRALA
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Diabetis; Retinal Neovascularization; laser treatment
MeSH Terms: conditions — Retinal Neovascularization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SS-PRP arm (Active Comparator): panfotocoagulation (PRP) single shoot (ETDRS) + 0,05ml intravitreal injection anti-VEGF (ranibizumabe)
  Interventions: Drug: Intravitreal Ranibizumabe; Drug: panfotocoagulation (PRP) single shoot (ETDRS)
- MS-PRP arm (Experimental): Multiple shoot panfotocoagulation (PASCAL) plus IVR
  Interventions: Drug: Intravitreal Ranibizumabe; Drug: panfotocoagulation (PASCAL)
- IVR arm (Other): only IVR (intravitreal Ranibizumabe)
  Interventions: Drug: Intravitreal Ranibizumabe

INTERVENTIONS:
Drug: Intravitreal Ranibizumabe — Intravitreal injection 0,05ml Ranibizumabe
Drug: panfotocoagulation (PASCAL)
  Arms: MS-PRP arm
Drug: panfotocoagulation (PRP) single shoot (ETDRS)
  Arms: SS-PRP arm

SUMMARY:
Objectives:

Primary objective:

To evaluate the effects on retinal morphophysiology of full scatter single target panretinal photocoagulation (PRP) versus full scatter multiple target panretinal photocoagulation (both combined with intravitreous injections of ranibizumab) versus intravitreous ranibizumab (IVR) alone in patients with proliferative diabetic retinopathy (PDR).

Primary outcome:

The primary endpoint for this study is the mean change in the total area of active retinal neovessels, as measured by fluorescein angiography leakage area, in mm2, from baseline to week 48.

Secondary objectives:

* To assess the mean changes in best corrected visual acuity (BCVA), the mean changes in central subfield foveal thickness (CSFT), the mean changes in wave B amplitude and oscillatory potentials on a full-field electroretinogram (ERG), and the mean changes on the peripheral visual field by static perimetry (30:2 strategy), from baseline to week 48.
* To assess the incidence of adverse events during the study.

Strategic goal:

In the era of anti-VEGF treatment for retinal neovascularization 1, 2, 3, 4 , it is time to determine what would be the best association of PRP + anti-VEGF for proliferative diabetic retinopathy (PDR), or still, if just intravitreal anti-VEGF treatment would be even better regarding morphologic (new vessels area and CSFT) and functional parameters (BCVA, ERG response and visual field).

DETAILED DESCRIPTION:
Photocoagulation (thermal laser) was the first modality to be described for the treatment of PDR. Different types of laser such as xenon, krypton, argon, red diode and green diode can be used for this treatment. The Early Treatment Diabetic Retinopathy Study (ETDRS) showed the benefit of early treatment of PDR and of macular edema with laser photocoagulation.

However, several studies have reported loss of visual field after laser photocoagulation of the bilateral full-scatter type (PRP) due to the expansion of the thermal injury, possibly even compromising the ability to drive automotive vehicles according to the standards of the transit authorities of some countries. Thus, this implies a greater impact on the quality of life of the patient, especially if he is a young diabetic.6

The objective of new laser photocoagulation technologies is to provide a treatment that will permit the development of a regenerative response of photoreceptors and of the retinal pigment epithelium (RPE) with the minimum loss of photoreceptors and the minimum cicatricial expansion of the thermal injury on the targeted RPE.7

The PASCAL photocoagulator (OptiMedica, Santa Clara, California) (a standard scanning laser) was introduced in 2005 for retinal photocoagulation. The device functions as if it partially automated the procedure by means of a shorter laser pulse (short pulse strategy) combined with multiple simultaneous firings in a pattern, performing the procedure within a shorter period of time and with less damage to the outer retina or the RPE, in addition to providing better patient comfort.8

Regarding combined therapy, the combination of intravitreous injection of ranibizumab with PRP (ETDRS) proved to be more promising in terms of improved visual acuity, stability of macular thickness and a greater regression rate of neovessel areas than the use of PRP alone (ETDRS) in patients with high risk PDR.1

Thus, in the present study we would like to determine which would be the best therapeutic combination of laser and an anti-VEGF drug for our patients, or whether treatment with an anti-VEGF drug alone would be better in terms of the anatomical and functional parameters proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic patients older than 18 years
2. Presence of PDR (presence of retinal neovascularization, defined as active neovessels (fine retinal vessels with saccular dilatations or extremities covered with blood or associated with recurrent vitreous hemorrhage) with visual acuity better than 20/800 and with no previous laser treatment
3. Giving written informed consent.

Exclusion Criteria:

1. Presence of advanced PDR, i.e.: vitreous hemorrhage that would prevent documentation of the eye fundus or adequate retinal photocoagulation, or presence of traction retinal detachment
2. Presence of ring-shaped retinal neovascularization extending along both temporal arcades and the optic disc
3. Any abnormality of the vitreoretinal interface in the macular region for which the investigator would consider vitrectomy via pars plana to be necessary
4. Intravitreous injection of corticosteroids or of other antiangiogenic drugs 6 months before the evaluation for entry into the study
5. Inability to fixate and to conclude the automated static perimetry exam
6. Cataract surgery within the last three months
7. Posterior vitrectomy with scleral introflexion at any time
8. Acute ocular infection
9. Allerghy to fluorescein
10. Medical or psychological conditions that would prevent the patient from giving informed consent and concluding the study
11. Significant uncontrolled diseases which, in the opinion of the investigator, would exclude the patient from the study
12. Renal failure requiring dialysis or renal transplant or renal insufficiency with creatinine levels >2.0 mg/dl
13. Untreated diabetes mellitus
14. Severe (blood pressure systolic > 160 mmHg or diastolic > 100 mmHg) AND untreated hypertension
15. Inability to comply with study or follow-up procedures.
16. Impaired or limited legal capacity
17. Participation in another clinical study in the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
fluorescein angiography leakage area | from baseline to week 48.
  The primary endpoint for this study is the mean change in the total area of active retinal neovessels, as measured by fluorescein angiography leakage area, in mm2.

CONTACTS AND LOCATIONS:
Locations (1):
- Retina and Vitreous service of the University Hospital, Faculty of Medicine of Ribeirão Preto-USP (HCFMRP), Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Barroso RMP, Messias K, Garcia DM, Cardillo JA, Scott IU, Messias A, Jorge R. ETDRS panretinal photocoagulation combined with intravitreal ranibizumab versus PASCAL panretinal photocoagulation with intravitreal ranibizumab versus intravitreal ranibizumab alone for the treatment of proliferative diabetic retinopathy. Arq Bras Oftalmol. 2020 Nov-Dec;83(6):526-534. doi: 10.5935/0004-2749.20200096. PMID 33470281